CLINICAL TRIAL: NCT05599009
Title: Remote Ischemic Conditioning and Dynamic Cerebral Autoregulation in Patients With Intracranial and Extracranial Arteriosclerosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RIC-DCAS
Record Dates: First submitted 2022-10-10; First posted 2022-10-31 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2022-10

CONDITIONS: Carotid Stenosis; Ischemic Stroke
MeSH Terms: conditions — Carotid Stenosis; Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RIC group (Experimental): RIC+Standard medical treatment. Remote ischemic conditioning (RIC) is induced by 4 cycles of 5 min of healthy upper limb ischemia followed by 5 min re-perfusion. Limb ischemia was induced by inflation of a blood pressure cuff to 200 mmHg.
  Interventions: Procedure: remote ischemic conditioning
- control group (Sham Comparator): Sham RIC+Standard medical treatment. Sham remote ischemic conditioning (RIC) is induced by 4 cycles of 5 min of healthy upper limb ischemia followed by 5 min re-perfusion. Limb ischemia was induced by inflation of a blood pressure cuff to 60 mmHg.
  Interventions: Procedure: sham remote ischemic conditioning

INTERVENTIONS:
Procedure: remote ischemic conditioning — Remote ischemic conditioning (RIC) is induced by 4 cycles of 5 min of healthy upper limb ischemia followed by 5 min re-perfusion. Limb ischemia was induced by inflation of a blood pressure cuff to 200 mmHg. All patients underwent dynamic cerebral autoregulation before treatment, immediately after treatment, 6 hours after treatment and 24 hours after treatment.
  Arms: RIC group
Procedure: sham remote ischemic conditioning — Remote ischemic conditioning (RIC) is induced by 4 cycles of 5 min of healthy upper limb ischemia followed by 5 min re-perfusion. Limb ischemia was induced by inflation of a blood pressure cuff to 60 mmHg. All patients underwent dynamic cerebral autoregulation before treatment, immediately after treatment, 6 hours after treatment and 24 hours after treatment.
  Arms: control group

SUMMARY:
The purpose of this study is to explore the effect of remote ischemic conditioning on the dynamic cerebral autoregulation in patients with intracranial and extracranial arteriosclerosis and the changes of dynamic cerebral autoregulation within 24 hours after remote ischemic conditioning.

DETAILED DESCRIPTION:
In this study, patients with intracranial and extracranial arteriosclerosis were included. The experimental group received basic treatment and remote ischemic conditioning for 200mmHg to pressurize the upper arm of the healthy side for 5 minutes, relax for 5 minutes, and repeat 4 cycles. The control group received basic treatment and remote ischemic conditioning for 60mmHg to pressurize the upper arm of the healthy side for 5 minutes, relax for 5 minutes, and repeat 4 cycles. The dynamic cerebral autoregulation was measured before treatment, immediately after treatment, 6 hours after treatment and 24 hours after treatment in both groups. The investigators aimed to determine the effect of remote ischemic conditioning on the dynamic cerebral autoregulation in patients with intracranial and extracranial arteriosclerosis. The investigators hypothesized that remote ischemic conditioning would improve dynamic cerebral autoregulation in patients with intracranial and extracranial arteriosclerosis.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥18 years, < 80 years, regardless of sex;
2. Patients with clinically definite diagnosis of intracranial and extracranial atherosclerosis.
3. Baseline Glasgow Coma Scale (GCS) ≥8;
4. Be able to accept remote ischemic conditioning;
5. Bilateral temporal windows were well penetrated;
6. Signed and dated informed consent is obtained

Exclusion Criteria:

1. Patients who undergo intravenous thrombolysis or endovascular treatment;
2. Patients with consciousness disorder or restlessness who cannot cooperate with dynamic cerebral autoregulation;
3. Patients whose stable cerebral blood flow velocity envelope cannot be obtained by transcranial Doppler ultrasound or whose cerebral blood vessels have not been detected;
4. Patients with severe arrhythmia (frequent ventricular or supraventricular arrhythmia diagnosed by 24 hours dynamic ECG), hyperthyroidism, severe anemia, unstable blood pressure and other factors affecting the hemodynamics;
5. CT shows cerebral hemorrhagic diseases: hemorrhagic stroke, epidural hematoma, subdural hematoma, intracranial hematoma, ventricular hemorrhage, subarachnoid hemorrhage, etc;
6. Other intracranial lesions, such as cerebrovascular malformations, cerebral venous lesions, tumors and other diseases involving the brain craniocerebral planning for surgical treatment;
7. Other serious diseases and have a life expectancy of less than 3 months;
8. Serious blood system diseases or severe coagulation dysfunction;
9. Severe organ dysfunction or failure;
10. Previously received remote ischemic conditioning or similar treatment;
11. Contraindications of remote ischemic conditioning, such as severe soft tissue injury, fracture or vascular injury, peripheral vascular disease in the contralateral upper limb;
12. Unqualified laboratory test indicators: Aspartate aminotransferase or alanine aminotransferase was 3 times higher than the upper limit of normal range, serum creatinine was > 265umol/l (> 3mg/dl), platelet was < 100×109/ l, international normalized ratio (INR), activated partial thromboplastin time (APTT), prothrombin time (PT) were above the upper limit of normal range;
13. Pregnant or lactating women;
14. Participating in other clinical investigators, or having participated in other clinical investigators within 3 months before enrollment;
15. Patients who do not follow up or have poor treatment compliance;
16. Other conditions deemed inappropriate for inclusion by the investigator

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2022-12-10 (Actual); Primary Completion 2023-02-28 (Estimated); Study Completion 2023-02-28 (Estimated)

PRIMARY OUTCOMES:
Dynamic cerebral autoregulation parameters (PD) | 0-6 hours
  Dynamic brain autoregulation parameters obtained from transfer function analysis in degrees. Continuous cerebral blood flow velocities of bilateral middle cerebral artery will be assessed noninvasively using transcranial Doppler. Spontaneous arterial blood pressure will be simultaneously recorded using a servo-controlled plethysmograph on the left or right middle finger with an appropriate finger cuff size. Transfer function analysis will be used to derive the autoregulatory parameters.

SECONDARY OUTCOMES:
Dynamic cerebral autoregulation parameters (PD) | 0-1 hours
  Dynamic brain autoregulation parameters obtained from transfer function analysis in degrees. Continuous cerebral blood flow velocities of bilateral middle cerebral artery will be assessed noninvasively using transcranial Doppler. Spontaneous arterial blood pressure will be simultaneously recorded using a servo-controlled plethysmograph on the left or right middle finger with an appropriate finger cuff size. Transfer function analysis will be used to derive the autoregulatory parameters.
Dynamic cerebral autoregulation parameters (PD) | 0-24 hours
  Dynamic brain autoregulation parameters obtained from transfer function analysis in degrees. Continuous cerebral blood flow velocities of bilateral middle cerebral artery will be assessed noninvasively using transcranial Doppler. Spontaneous arterial blood pressure will be simultaneously recorded using a servo-controlled plethysmograph on the left or right middle finger with an appropriate finger cuff size. Transfer function analysis will be used to derive the autoregulatory parameters.

CONTACTS AND LOCATIONS:
Locations (1):
- First Hospital of Jilin University, Changchun, Jilin, China